CLINICAL TRIAL: NCT05877287
Title: The Effect of Mındfulness-Based Stress Reductıon Program Applıed to Parents Wıth A Chıld Wıth Autısm on The Level Of Depressıon, Anxıety, Stress and Hopelessness: Randomızed Controlled Trıal
Brief Title: Effect of Awareness-Based Stress Reducatıon Program Applıed to Parents Wıth A Chıld Wıth Autısm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Selverhan Yurttutan, RESEARCH ASSISTANT, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/410:13610
Record Dates: First submitted 2023-05-15; First posted 2023-05-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: DEPRESSION; ANXIETY; STRESS; HOPELESSNESS; MİNDFULNESS
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: parallel group (experiment-control) randomized controlled experimental
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based stress reduction program (Experimental): The FTSA program will be carried out once a week for 60 minutes, for 8 weeks, in a total of 8 sessions. The program will be conducted in face-to-face groups. Sessions will be held in a suitable area in the practice area. In each 60-minute session, it is planned to be 20 minutes of narration on the subject of the session, accompanied by a power point presentation, and the remaining 40 minutes of exercise, meditation practices and sharing experiences.
  Interventions: Other: mindfulness-based stress reduction program
- control group (No Intervention): No application will be made.

INTERVENTIONS:
Other: mindfulness-based stress reduction program — The FTSA program will be carried out once a week for 60 minutes, for 8 weeks, in a total of 8 sessions. The program will be conducted in face-to-face groups. Sessions will be held in a suitable area in the practice area. In each 60-minute session, it is planned to be 20 minutes of narration on the subject of the session, accompanied by a power point presentation, and the remaining 40 minutes of exercise, meditation practices and sharing experiences.
  Arms: mindfulness-based stress reduction program

SUMMARY:
This research was planned to examine the effect of mindfulness-based stress reduction program applied to parents with autistic children on the level of depression, anxiety, stress and hopelessness.

DETAILED DESCRIPTION:
The program applied to parents with children with autism will be carried out once a week for 60 minutes, for 8 weeks, in 8 sessions in total. The program will be conducted in face-to-face groups. Sessions will be held in a suitable area in the practice area. In each 60-minute session, it is planned to be 20 minutes of narration on the subject of the session, accompanied by a power point presentation, and the remaining 40 minutes of exercise, meditation practices and sharing experiences. In the table indicating the general operation of the sessions within the scope of the research; The purpose, target, teaching method, material place, time, session content and application steps of each session will be given to the participants. Awareness-Based Stress Reduction Program Applied to Parents with Children with Autism will be given to the participants in the first week, including the important points of the program, prepared by the researchers, and expert opinions will be taken.

ELIGIBILITY:
Inclusion Criteria

* Being a parent of a child with autism
* Being literate and able to communicate in Turkish

Exclusion Criteria:

* Having a diagnosed mental and mental health problem
* Having a chronic, mental and mental health problem other than autism in a child with autism
* Having previously participated in a mindfulness-based stress reduction program
* Having another disabled child

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale (DASS-21) | First assessment will be made at the baseline (pre-intervention)
  The scale consists of 21 items and three sub-dimensions. Each of the seven items that make up each sub-dimension of the scale measures depression, anxiety and stress. The DASS-21 scale is a four-point Likert-type scale and the items are evaluated between 0 and 3 (0 = not at all suitable for me, 1 = somewhat appropriate for me, 2 = usually suitable for me, 3 = completely suitable for me). There is no reverse item in the scale. The total scores of the scale range from 0 to 21 for each sub-dimension. In the validity and reliability study, the Cronbach-alpha coefficient was determined as 0.87 for the depression sub-dimension, 0.85 for the anxiety sub-dimension, and 0.81 for the stress sub-dimension. The Cronbach-alpha coefficient for the Turkish version of the Depression, Anxiety and Stress scale was determined as 0.88 for the depression sub-dimension, 0.80 for the anxiety sub-dimension and 0.87 for the stress sub-dimension (Sarıçam, 2018).
Depression, Anxiety and Stress Scale (DASS-21) | The second assessment will take place 8 weeks after the first assessment (after the program is completed).
  The scale consists of 21 items and three sub-dimensions. Each of the seven items that make up each sub-dimension of the scale measures depression, anxiety and stress. The DASS-21 scale is a four-point Likert-type scale and the items are evaluated between 0 and 3 (0 = not at all suitable for me, 1 = somewhat appropriate for me, 2 = usually suitable for me, 3 = completely suitable for me). There is no reverse item in the scale. The total scores of the scale range from 0 to 21 for each sub-dimension. In the validity and reliability study, the Cronbach-alpha coefficient was determined as 0.87 for the depression sub-dimension, 0.85 for the anxiety sub-dimension, and 0.81 for the stress sub-dimension. The Cronbach-alpha coefficient for the Turkish version of the Depression, Anxiety and Stress scale was determined as 0.88 for the depression sub-dimension, 0.80 for the anxiety sub-dimension and 0.87 for the stress sub-dimension (Sarıçam, 2018).
Depression, Anxiety and Stress Scale (DASS-21) | Third assessment will take place average 4 weeks after the second assessment.
  The scale consists of 21 items and three sub-dimensions. Each of the seven items that make up each sub-dimension of the scale measures depression, anxiety and stress. The DASS-21 scale is a four-point Likert-type scale and the items are evaluated between 0 and 3 (0 = not at all suitable for me, 1 = somewhat appropriate for me, 2 = usually suitable for me, 3 = completely suitable for me). There is no reverse item in the scale. The total scores of the scale range from 0 to 21 for each sub-dimension. In the validity and reliability study, the Cronbach-alpha coefficient was determined as 0.87 for the depression sub-dimension, 0.85 for the anxiety sub-dimension, and 0.81 for the stress sub-dimension. The Cronbach-alpha coefficient for the Turkish version of the Depression, Anxiety and Stress scale was determined as 0.88 for the depression sub-dimension, 0.80 for the anxiety sub-dimension and 0.87 for the stress sub-dimension (Sarıçam, 2018).

SECONDARY OUTCOMES:
Beck Hopelessness Scale (BUS) | First assessment will be made at the baseline (pre-intervention)
  It was developed to determine the degree of pessimism of the individual for the future. The scale, which consists of a total of 20 items, is scored between 0-1 and is a self-assessment type scale. It can also be applied as a group. It is a scale that can be easily applied to literate children, young people and adults without time limit. The scale is evaluated in three sub-dimensions regarding the future (Future Emotions, Loss of Motivation, Future Expectations). 20 items in the scale are answered as "Yes and No", each inconsistent answer is scored with 0 and each compatible answer with 1 point. "yes" to eleven items (2, 4, 7, 9, 11, 12, 14, 16, 17, 18, 20) and 9 items (1, 3, 5, 6, 8, 10, 13, 15, 19) "no" answer is evaluated with 1 point. A high total score (in the range of 0-20) is considered as "high level of hopelessness".
Beck Hopelessness Scale (BUS) | The second assessment will take place 8 weeks after the first assessment (after the program is completed).
  It was developed to determine the degree of pessimism of the individual for the future. The scale, which consists of a total of 20 items, is scored between 0-1 and is a self-assessment type scale. It can also be applied as a group. It is a scale that can be easily applied to literate children, young people and adults without time limit. The scale is evaluated in three sub-dimensions regarding the future (Future Emotions, Loss of Motivation, Future Expectations). 20 items in the scale are answered as "Yes and No", each inconsistent answer is scored with 0 and each compatible answer with 1 point. "yes" to eleven items (2, 4, 7, 9, 11, 12, 14, 16, 17, 18, 20) and 9 items (1, 3, 5, 6, 8, 10, 13, 15, 19) "no" answer is evaluated with 1 point. A high total score (in the range of 0-20) is considered as "high level of hopelessness".
Beck Hopelessness Scale (BUS) | Third assessment will take place average 4 weeks after the second assessment.
  It was developed to determine the degree of pessimism of the individual for the future. The scale, which consists of a total of 20 items, is scored between 0-1 and is a self-assessment type scale. It can also be applied as a group. It is a scale that can be easily applied to literate children, young people and adults without time limit. The scale is evaluated in three sub-dimensions regarding the future (Future Emotions, Loss of Motivation, Future Expectations). 20 items in the scale are answered as "Yes and No", each inconsistent answer is scored with 0 and each compatible answer with 1 point. "yes" to eleven items (2, 4, 7, 9, 11, 12, 14, 16, 17, 18, 20) and 9 items (1, 3, 5, 6, 8, 10, 13, 15, 19) "no" answer is evaluated with 1 point. A high total score (in the range of 0-20) is considered as "high level of hopelessness".

CONTACTS AND LOCATIONS:
Overall Officials: Emine GEÇKİL, Prof. Dr., Study Director — Necmettin Erbakan Univercity
Locations (1):
- Necmettin Erbakan Üniversity, Konya, Turkey (Türkiye)